CLINICAL TRIAL: NCT06924905
Title: Exploring Pelvic Floor Dysfunction Among Egyptian Female Athletes: Prevalence, Risk Factors, and Implications for Performance
Brief Title: Exploring Pelvic Floor Dysfunction Among Egyptian Female Athletes
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, director of scientific committee, Cairo University
Other Study IDs: P.T.REC/012/005380
Record Dates: First submitted 2025-04-05; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Sports; Public Health; Female; Pelvic Diseases
Keywords: Public Health; Pelvic Disorders; pelvic dysfunctions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: the pelvic floor disability index — 20 questions divided into three sections: Pelvic Organ prolapse Distress Inventory 6 (POPDI-6), Colorectal-Anal distress Inventory 8 (CRAD-8) and Urinary distress Inventory 6 (UDI-6).

SUMMARY:
This Study is aiming to identify the prevalence of pelvic floor dysfunction in female athletes in Egypt and which sports contribute more in increasing their number. helping in gathering information about the risk factors and raising awarness about Pelvic floor dysfunction

DETAILED DESCRIPTION:
RESEARCH QUESTION:

Is there high prevalence of pelvic floor dysfunction among athletic females in Egypt and if there is specific sports contributing to that? the Sample are the Females recruited from different clubs across Egypt, female athletes who participated in previous studies and got thier contact and consent and by a Google form sent via links through social media aiming to reach a wide varieties of athletes across egypt . They will be selected according to the following eligibility criteria. the pelvic floor disability index will be used to evaluate pelvic floor. The questionnaire, transferred to Google Form, consists of 20 questions divided into three sections: Pelvic Organ prolapse Distress Inventory 6 (POPDI-6), Colorectal-Anal distress Inventory 8 (CRAD-8) and Urinary distress Inventory 6 (UDI-6). Fifteen participants, randomly selected by administrative staff, academics, and students of the Faculty of Physiotherapy at Cairo University, will test the questionnaire to identify any issues with language or format.

Data will be analyzed using IBM SPSS (version 22) for Windows. Demographic data will be analyzed using ANOVA. Bivariate correlation will be used to assess relationships between pelvic floor dysfunction and risk factors and demographic data. A p-value less than 0.05 will be considered statistically significant.

our criteria consists of

Inclusion Criteria:

* Their age will range from 16 to 60 years.
* Female gender only.
* Females engaged in regular sports or athletic activities..
* Currently residing in Egypt

Exclusion Criteria:

* Not currently involved in sports or physical activities.
* Egyptian females living outside Egypt.
* Participants involved in para-athletics. the concent from the participants is taken either verbally or Via the google form sent as mentioned above there will be a consent declaration at the beginning of the form for the participants to approve to participate.

as for the participant withdrawl : A thorough description of the procedure will be explained and they understand they may withdraw their consent and discontinue participation in this research and no consequences for the participant in withdrawing. Their data will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 16 to 60 years.
* Female gender only.
* Females engaged in regular sports or athletic activities..
* Currently residing in Egypt

Exclusion Criteria:

* Not currently involved in sports or physical activities.
* Egyptian females living outside Egypt.
* Participants involved in para-athletics.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females recruited from different clubs across Egypt
Study Population: Females recruited from different clubs across Egypt
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
pelvic floor disability index | 2 months
  the pelvic floor disability index will be used to evaluate pelvic floor. The questionnaire, transferred to Google Form, consists of 20 questions divided into three sections: Pelvic Organ prolapse Distress Inventory 6 (POPDI-6), Colorectal-Anal distress Inventory 8 (CRAD-8) and Urinary distress Inventory 6 (UDI-6).